CLINICAL TRIAL: NCT04018833
Title: Intravitreal Ranibizumab or Aflibercept After Bevacizumab in Diabetic Macular Edema
Acronym: SWITCH
Status: Completed | Type: Observational
Sponsor: Bernardete Pessoa MD (Other)
Responsible Party: Sponsor-Investigator, Bernardete Pessoa MD, Ophthalmologist, Centro Hospitalar do Porto
Organization: Centro Hospitalar do Porto (Other)
Other Study IDs: 20190701245703984
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: Diabetic Macular Edema; Bevacizumab; Ranibizumab; Aflibercept; BCVA; OCT
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ranibizumab: Patients nonresponsive to bevacizumab that were switched to ranibizumab
  Interventions: Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution [LUCENTIS]
- aflibercept: Patients nonresponsive to bevacizumab that were switched to aflibercept
  Interventions: Drug: Aflibercept 40 MG/ML Intraocular Solution [EYLEA]

INTERVENTIONS:
Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution [LUCENTIS]
  Groups: ranibizumab
Drug: Aflibercept 40 MG/ML Intraocular Solution [EYLEA]
  Groups: aflibercept

SUMMARY:
PURPOSE: To evaluate the efﬁcacy of switching from bevacizumab to ranibizumab (Lucentis; Genentech, South San Francisco, CA) or aflibercept (Eylea; Regeneron, Tarrytown, NY) in eyes with diabetic macular edema (DME) nonresponders to bevacizumab (Avastin; Genentech, South San Francisco, CA).

METHODS: Single-center retrospective comparative study of patients with DME unresponsive to intravitreal bevacizumab that were switched to ranibizumab or aflibercept. Best-corrected visual acuity and central foveal thickness will be analysed prior to and 3 months after the switch. OCT biomarkers will also analyzed.

A p value of 0.05 or less will be considered to be statistically significant. HYPOTHESIS: Patients will improve anatomically and functionally after switch.

ELIGIBILITY:
Inclusion Criteria:

* type 1 or type 2 diabetes mellitus patients
* older than 18 years
* with center-involved DME, defined as central subfield thickness (CST) of more than 300 µm on spectral-domain OCT (SD-OCT).
* nonresponsive to bevacizumab, deﬁned as having persistent intraretinal and/or subretinal fluid on optical coherence tomography (OCT), i.e CSF>300µm after a minimum of 3 monthly injections, 4 months before switch, regardless of visual acuity (VA).

Exclusion Criteria:

* additional ocular diseases that could significantly affect the visual acuity such as:
* significant vitreoretinal interface abnormality on SD-OCT that may contribute to macular edema
* age-related macular degeneration
* retinal vascular occlusion
* central corneal opacity
* amblyopia
* advanced glaucoma
* optic neuropathy
* history of ocular trauma or surgery other than uncomplicated cataract extraction
* cataract surgery within 3 months before or after bevacizumab switch
* unable to provide written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients followed on the ocular diabetes consultation of Centro Hospitalar Universitário do Porto, Portugal, with DME unresponsive or incompletly responsive to intravitreal bevacizumab (1,25 MG/0.05 ML).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Anatomical change | Immediately before switch (one month after last bevacizumab intravitreal injection); 4 months after switch. Minimum of three intravitreal injections before and after switch.
  The central foveal thickness (CFT), measured by Optical Coherence Tomography, was automatically measured by the software in the central 1 mm. A CFT <250 µm or >300 µm is considered pathological. A CFT between 200 and 300 µm is considered physiological. CFT has no defined minimum or maximum values.
  Since patients with diabetic macular edema usually have CFT >300 µm the goal of treatment is to lower the CFT to values between 200 and 300 µm. A clinical significant anatomical improvement was considered for a change in CFT≥10%.
Functional change | Immediately before switch (one month after last bevacizumab intravitreal injection); 4 months after switch. Minimum of three intravitreal injections before and after switch.
  Functional change was measure by the Early Treatment Diabetic Retinopathy Scale (ETDRS) which measures the best-corrected visual acuity with an ETDRS-like chart at 4 meters in number letters or at 1 meter when patients are unable to read any letters on the ETDRS chart at 4 meters. The ETDRS scale varies from 1 to 85 letters (85 letters correspond to a 20/20 in the Snellen scale).
  The higher the value the better the outcome. A clinical significant functional improvement was considered for a gain of ≥5 EDTRS letters.

CONTACTS AND LOCATIONS:
Overall Officials: João Melo-Beirão, MD, PhD, Study Director — Centro Hospitalar do Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pessoa B, Malheiro L, Carneiro I, Monteiro S, Coelho J, Coelho C, Figueira J, Meireles A, Melo Beirao JN. Intravitreal Ranibizumab or Aflibercept After Bevacizumab in Diabetic Macular Edema: Exploratory Retrospective Analysis. Clin Ophthalmol. 2021 Jan 22;15:253-260. doi: 10.2147/OPTH.S280644. eCollection 2021. PMID 33519187